CLINICAL TRIAL: NCT07237061
Title: Patient-preferred Aromatherapy Versus Placebo For Reducing Preoperative Anxiety In Patients Undergoing Eye Surgery - The RELAAC Randomised Controlled Trial
Brief Title: Patient-preferred Aromatherapy Versus Placebo For Reducing Preoperative Anxiety In Patients Undergoing Eye Surgery
Acronym: RELAAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2020/01202
Record Dates: First submitted 2025-06-26; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-06

CONDITIONS: Cataract; Surgery; Vitrectomy; Aromatherapy; Preoperative Anxiety
Keywords: randomized controlled trial; placebo controlled; double blinded; two arm
MeSH Terms: conditions — Cataract | interventions — Aromatherapy; lavender oil; lemongrass oil

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- placebo (Placebo Comparator): Patients were asked to choose amongst 4 different aromatherapy scents. The study administrator then stuck an adhesive patch without any aromatherapy oil on it, to the patient's facemask. This was worn throughout the perioperative experience from the ambulatory ward to the operating theatre and post anaesthesia care unit (PACU).
  Interventions: Other: Placebo
- intervention (Experimental): Patients were asked to choose amongst 4 different aromatherapy scents. The study administrator then stuck an adhesive patch with 1 drop of their chosen aromatherapy oil on it, to the patient's facemask. This was worn throughout the perioperative experience from the ambulatory ward to the operating theatre and post anaesthesia care unit (PACU).
  Interventions: Other: Aromatherapy

INTERVENTIONS:
Other: Aromatherapy — patients chose their preferred aromatherapy scent to be used for at least 30 minutes
  Other Names: lavender; geranium; lemongrass; sandalwood
  Arms: intervention
Other: Placebo — odorless dry absorbent adhesive patch
  Arms: placebo

SUMMARY:
This study looks at whether aromatherapy (scent chosen by the patient), is better than routine care, at reducing preoperative anxiety before eye surgery.

ELIGIBILITY:
Inclusion Criteria:

* mental capacity for informed consent
* undergoing elective ambulatory eye surgery (including Phacoemulsification, Femtosecond laser-assisted cataract surgery (FLACS), Extracapsular cataract extraction (ECCE) and vitrectomy).
* surgery only under Monitored Anaesthesia Care (MAC)3
* surgical duration less than 45 minutes

Exclusion Criteria:

* anosmia
* allergy to aromatherapy oil
* asthma
* allergic rhinitis
* psychiatric disease
* altered mental state
* lack of mental capacity
* active infection
* pregnancy
* patient or surgeon refused participation

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
change in VAS scores for preoperative anxiety | 30-60 minutes
  preoperative anxiety was ranked by the patient on a scale of 0-100 on a visual acuity scale (VAS) measuring 100mm, in the preoperative ambulatory ward, before and after the intervention/placebo was applied for at least 30 minutes. The change in the VAS score at these 2 timepoints was the primary outcome

CONTACTS AND LOCATIONS:
Locations (1):
- National University Hospital Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
local Patient Data Protection Act